CLINICAL TRIAL: NCT01367704
Title: A Randomized Controlled Trial of an Adolescent Relationship Abuse Prevention Program Entitled "Coaching Boys Into Men"
Brief Title: Evaluation Of "Coaching Boys Into Men" (CBIM) Program
Acronym: CBIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Miller, Chief, Division of Adolescent Medicine, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO11060186; 1R01CE001561-01 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Violence; Abuse
Keywords: gender-based violence; intimate partner violence; relationship abuse; sexual harassment; sexual violence
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control School (Active Comparator): Control schools (where the coaches do not receive the Coaching Boys into Men (CBIM) training until following academic year 'wait list control')
  Interventions: Behavioral: "Coaching Boys Into Men" program
- Intervention School (Experimental): Intervention schools (where coaches receive the CBIM training at start of sports season)
  Interventions: Behavioral: "Coaching Boys Into Men" program

INTERVENTIONS:
Behavioral: "Coaching Boys Into Men" program — Coaching Boys into Men (CBIM) program consists of a 60 minute training for high school coaches led by a violence prevention advocate to introduce coaches to the rationale for CBIM and the CBIM Coaches Kit. The Coaches use this CBIM toolkit to provide weekly discussions with their athletes (generally 10-15 minute mini-sessions) throughout their athletic season (11 weeks). Discussion topics include how to prevent disrespectful and harmful behaviors towards women and girls and how to promote healthy choices and relationships among youth.

SUMMARY:
Despite the high prevalence of adolescent relationship abuse (ARA) reported among adolescent females and substantial reports of perpetration by young males, effective prevention programs to prevent ARA are limited. Male athletes are an important target for prevention efforts given their higher rates of abuse perpetration compared to non-athlete peers as well as their social influence among their peers. This cluster-randomized school-based investigation examines the effectiveness of a program for the primary prevention of ARA. "Coaching Boys into Men" (CBIM) is a social norms theory-based program intended to alter norms that foster ARA perpetration, promote bystander intervention, and reduce ARA perpetration by engaging athletic coaches as positive role models to deliver violence prevention scripts and tools to high school age male athletes. Coaches receive a 60-minute training session to administer the intervention to their athletes via 11 lessons across a sport season. Trained high school coaches talk to their male athletes about 1) what constitutes disrespectful and harmful vs. respectful behaviors, 2) promoting more gender-equitable attitudes, and 3) modeling bystander intervention when disrespectful behaviors toward women and girls are witnessed. The current investigation evaluates the intervention in 16 urban high schools randomized either to receive the CBIM program (i.e., intervention schools, n=8) or to a control condition (n=8). Baseline computer-based surveys are collected for all intervention and control site student athletes entering grades 9 through 12 at the start of each of three sports seasons across Year 1 (Time 1). Follow up surveys are collected for these same athletes at the end of their first sports season (Time 2). Participating athletes in grades 9 - 11 at baseline are re-surveyed 12 months after Time 1 to examine the longer term effects of the CBIM intervention (Time 3; N of athletes completing all 3 waves of data collection = 1500). Primary assessment of intervention effects are based on intent-to-treat estimates, utilizing generalized linear mixed models to account for clustering arising from school randomization. Hypothesized outcomes for male athletes include a) an increase in recognition of what constitutes abusive behaviors, b) more gender-equitable attitudes, c) an increase in intentions and reports of bystander intervention regarding ARA, and through these intermediate outcomes, d) a decrease in perpetration of ARA among adolescent male athletes.

DETAILED DESCRIPTION:
Additional process evaluation includes baseline and follow up surveys with coaches (from both intervention and control arms), individual interviews with coaches, as well as focus groups with students to collect coach and athlete perspectives on the relevance and local impact of the intervention program.

ELIGIBILITY:
School Eligibility:

Inclusion Criteria

-urban and suburban public high schools in Sacramento region with athletics program

Exclusion Criteria -private high schools, rural high schools

Coach Eligibility:

Inclusion Criteria

* coaching an athletic team at one of the participating schools (intervention or control)
* age 18 or older

Exclusion Criteria

-not coaching an athletic team at the participating schools

Athlete Eligibility:

Inclusion Criteria

* ages 14-18 (grades 9 to 12)
* student at one of the participating high schools
* able to read English
* participating in an athletic program led by a coach willing to participate in the research study

Exclusion Criteria

* outside age range
* not participating on sports team at the high school in which they are enrolled

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2006 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — Children's Hospital of Pittsburgh, University of Pittsburgh Medical Center
Locations (1):
- Children's Hospital of Pittsburgh, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jones KA, Tancredi DJ, Abebe KZ, Paglisotti T, Miller E. Cases of Sexual Assault Prevented in an Athletic Coach-Delivered Gender Violence Prevention Program. Prev Sci. 2021 May;22(4):504-508. doi: 10.1007/s11121-021-01210-1. Epub 2021 Jan 22. PMID 33481150
- [Derived] Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MCD, Anderson HA, O'Connor B, Silverman JG. One-year follow-up of a coach-delivered dating violence prevention program: a cluster randomized controlled trial. Am J Prev Med. 2013 Jul;45(1):108-112. doi: 10.1016/j.amepre.2013.03.007. PMID 23790995
- [Derived] Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MC, Anderson HA, Stetkevich N, Brown EW, Moideen F, Silverman JG. "Coaching boys into men": a cluster-randomized controlled trial of a dating violence prevention program. J Adolesc Health. 2012 Nov;51(5):431-8. doi: 10.1016/j.jadohealth.2012.01.018. Epub 2012 Mar 25. PMID 23084163

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control School | Intervention School
Started | 998 | 1008
Completed | 951 | 847
Not Completed | 47 | 161
Not completed — Lost to Follow-up | 47 | 161

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control School | Intervention School | Total
Number analyzed (Participants) | 998 | 1008 | 2006
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 998 | 1008 | 2006
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 998 | 1008 | 2006
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 998 | 1008 | 2006
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 169 | 220 | 389
  Not Hispanic or Latino | 822 | 776 | 1598
  Unknown or Not Reported | 7 | 12 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 114 | 78 | 192
  Native Hawaiian or Other Pacific Islander | 33 | 61 | 94
  Black or African American | 191 | 248 | 439
  White | 567 | 502 | 1069
  More than one race | 86 | 107 | 193
  Unknown or Not Reported | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 3 Months Using the Recognition of Abusive Behavior Scale
Description: Recognition of disrespectful and harmful behaviors against girls as abusive comparing baseline and follow up mean scores, using a 5-point Likert-like scale ranging from "not abusive" to "extremely abusive" (minimum = 1 and maximum = 5). This scale was developed by Silverman et al to assess perceptions of the degree of abusiveness of specified relationship behaviors and modeled as a mean of responses to 12 items.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mean scores
Arm/Group | Control School | Intervention School
Number analyzed (Participants) | 951 | 847
mean scores | 3.38 (.82) | 3.37 (.92)

2. Primary Outcome: Change From Baseline to 3 Months Using the Gender Equitable Attitudes Scale
Description: Assessment of gender-equitable attitudes comparing baseline mean score with follow up mean score, using a 5-point Likert-like scale ranging from "strongly agree" to "strongly disagree" (minimum = 1 and maximum = 5). This scale includes questions modified from Barker's Gender-Equitable Norms Scale and modeled as a mean of responses to 11 items.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mean scores
Arm/Group | Control School | Intervention School
Number analyzed (Participants) | 951 | 847
mean scores | 3.09 (.63) | 3.00 (.65)

3. Primary Outcome: Change From Baseline to 3 Months Using the Intentions to Intervene Scale
Description: Proclivity to intervene when witnessing disrespectful and harmful behaviors among peers comparing baseline and follow up mean scores, using a 5-point Likert-like scale ranging from "very unlikely" to "very likely" (minimum = 1 and maximum = 5). This scale was investigator developed by Miller (PI) et al to assess participants report of how likely they would be to do something to stop the behavior and modeled as a mean of 8 items.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mean scores
Arm/Group | Control School | Intervention School
Number analyzed (Participants) | 951 | 847
mean scores | 3.51 (.75) | 3.73 (.81)

ADVERSE EVENTS:
Arm/Group | Control School | Intervention School
Serious Adverse Events (participants affected / at risk) | 0/998 | 0/1008
Other Adverse Events (participants affected / at risk) | 0/998 | 0/1008

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No